CLINICAL TRIAL: NCT00779194
Title: Prospective Study of Rapamycin for the Treatment of SLE
Acronym: Rapamune
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Andras Perl, Professor of Medicine, Division Chief of Rheumatology, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#5658
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- SLE subjects (Experimental): SLE subjects receiving the study drug, Rapamune.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Rapamycin, is given to this group at a starting dose of 2 mg/day.
  Other Names: Rapamune; Sirolimus

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune disease of unknown origin. It involves multiple organs including the joints, skin, kidneys and central nervous system. The disease process is caused by a dysfunction of the immune system. The drugs currently used for the treatment of SLE are only partially effective and carry significant risks for side-effects. Patients that were resistant or intolerant to conventional medication have been effectively treated with Rapamycin and were able to decrease the amount of prednisone they needed.

The purpose of this study is to prospectively determine the therapeutic efficacy and mechanism of action of Rapamune in patients with SLE. Healthy subjects not receiving Rapamune will be asked to donate blood to serve as controls only for immunobiological outcomes.

As part of the research effort to understand the reason for the variations in the effects of treatment drugs by different individuals, a sub-study of the DNA makeup of subjects enrolled in the trial will also be done. The purpose of the sub-study is to possibly determine whether different responses to the drugs used to treat SLE have a correlation with the differences in the genetic makeup of the subjects.

DETAILED DESCRIPTION:
43 SLE subjects and 56 healthy controls are being recruited. The study will last 1 year with 9 study visits from day 0 to day 360. The healthy controls only need to donate blood once.

The study drug, sirolimus, is taken by mouth at a starting dose of 2mg/day. The dose is adjusted to achieve blood levels in the range of 6-15 ng/ml (the levels found to be effective for preventing organ rejections).

Blood samples are obtained before taking sirolimus, every two weeks for the first month, then every three months until 1 year, and then three months later to check the effect of discontinuing rapamycin. Each SLE subject will be asked to provide up to 100 ml (20 teaspoons) of blood at each visit. The first 6 visits will take place within 3 months and the remaining 3 visits every 3 months.

Routine laboratory work will be performed. Part of the blood drawn will be used for research and part will be used for routine lab work as part of standard of care.

The non-routine laboratory studies include:

1. Assessment of mitochondrial function in intact T cells
2. Analysis of mTOR activity, FKBP12 expression, and global gene expression in lupus T cells.
3. Predictors of therapeutic efficacy of sirolimus in SLE.

The study drug levels will be checked at every visit. The non-routine laboratory studies will be performed at Visits 0 and 8 for SLE subjects and at Visit 0 for the healthy control subjects.

Healthy control subjects will be matched by age (a decade or less), gender, and ethnic origin. They will be recruited and analyzed only for immunobiological outcomes on the same day as lupus subjects.

All subjects will sign an informed consent at visit 0. There is a separate informed consent for the main study, one for the SLE subjects and one for the Healthy Controls. The same subjects can participate in the genetic sub-study. They must sign another informed consent for the genetic sub-study, one for the SLE subjects and one for the Healthy Controls. There is no need for additional blood drawing since part of the blood drawn for the main study can be used for the genetic sub-study.

ELIGIBILITY:
Inclusion Criteria:

For SLE Subjects:

* SLE patients who exhibit ongoing disease activity by SLEDAI greater or equal to 4.
* SLE patients whose disease activity is controlled by administration of corticosteroids, most commonly, at least 10 mg/day of prednisone.
* 18 years of age or older.
* Updated vaccinations prior to study entry.
* Use of effective contraception for male patients before, during and up to 12 weeks after sirolimus therapy.

For Healthy Control Subjects:

* 18 years of age or older
* Must be matched with one of the SLE patients enrolled in the study by age, gender and ethnic origin
* Must not have any acute or chronic illness.

Exclusion Criteria:

For SLE Subjects:

* Patients who are pregnant.
* Patients with allergy or intolerance to sirolimus.
* Patients with life-threatening manifestations of SLE.
* Patients with proteinuria exceeding 500 mg/24 h or urine protein/creatine ratio >0.5.
* Patients with total cholesterol > 300 mg/dl or triglyceride > 400 mg.dl will be excluded.
* Patients with acute infection requiring antibiotics.
* Patients on sirolimus who develop infections and require intravenous antibiotics and fail to show clinical improvement in 5 days.
* Patients concurrently undergoing B cell-depleting therapy, cyclophosphamide, cyclosporine, and tacrolimus.
* Patients who have received investigational biologic B-cell depleting products within one year of study initiation.
* Patients with a history of chronic viral infections (e.g., HIV, hepatitis B, hepatitis C) or with a history of a malignancy (except non-melanoma skin cancer).
* Due to interference with sirolimus metabolism, subjects will not be allowed to receive concomitant rifampin, ketoconazole,voriconazole, itraconazole, erythromycin, or clarithromycin during the study.
* Patients with any type of interstitial lung disease.

For Healthy control Subjects:

* Subjects who are pregnant.
* Subjects with any acute or chronic illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Result] Lai ZW, Kelly R, Winans T, Marchena I, Shadakshari A, Yu J, Dawood M, Garcia R, Tily H, Francis L, Faraone SV, Phillips PE, Perl A. Sirolimus in patients with clinically active systemic lupus erythematosus resistant to, or intolerant of, conventional medications: a single-arm, open-label, phase 1/2 trial. Lancet. 2018 Mar 24;391(10126):1186-1196. doi: 10.1016/S0140-6736(18)30485-9. Epub 2018 Mar 15. PMID 29551338

RESULTS

PARTICIPANT FLOW:
Groups:
- SLE Subjects Receiving the Study Drug: SLE subjects receiving the study drug, Rapamune.
  Rapamycin: Rapamycin, is given to this group at a starting dose of 2 mg/day.
- Controls: Healthy control group donating blood only for immunobiological outcomes.
Period: Overall Study
Arm/Group | SLE Subjects Receiving the Study Drug | Controls
Started | 43 | 56
Completed | 29 | 56
Not Completed | 14 | 0

BASELINE CHARACTERISTICS:
Population: SLE patients and healthy controls (Blood samples of healthy individuals were obtained as controls only for immunobiological outcomes)
Groups:
- SLE Subjects Receiving the Study Drug: SLE Subjects Receiving the Study Drug, Rapamune. Rapamycin: Rapamycin, is given to this group at a starting dose of 2mg/day.
- Controls: Blood samples of healthy individuals were obtained as controls only for immunobiological outcomes.
- Total: Total of all reporting groups
Arm/Group | SLE Subjects Receiving the Study Drug | Controls | Total
Number analyzed (Participants) | 40 | 56 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 55 | 92
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14) | 45 (12) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 51 | 89
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 40 | 56 | 96

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Disease Activity as Measured by SLEDAI and BILAG Scores.
Description: The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) and The British Isles Lupus Assessment Group (BILAG) are clinical tools for assessing disease activity in lupus erythematosus patients. These indices play a central role as core determinants in SLE Responder Index.
  SLEDAI, comprising 24 items, quantifies disease activity on a scale of 0 to 105. Higher scores indicate more severe disease activity, reflecting cumulative impact of clinical and laboratory variables.
  BILAG, a comprehensive assessment, encompasses 97 items organized into 9 organ domains. The scoring ranges from A to E:
  A: No activity B: Mild activity C: Moderate activity D: Severe activity E: Very severe activity Total BILAG score is sum of individual item scores across all domains, with a potential range from 0 (if all items are graded as A, denoting no activity) to 97 (if all items are graded as E, signifying very severe activity). A lower total BILAG score indicates less severe disease activity.
Time Frame: 1 year
Population: SLE patients
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SLE Subjects Receiving the Study Drug: SLE subjects receiving the study drug Rapamune. Rapamycin: Rapamycin, is given to this group at a starting dose of 2 mg/day.
Arm/Group | SLE Subjects Receiving the Study Drug
Number analyzed (Participants) | 40
score on a scale
  SLEDAI | 10.2 (5.6)
  BILAG | 28.4 (12.4)

2. Secondary Outcome: Decrease of the Amount of Prednisone Needed to Control Disease Activity in SLE Patients.
Description: Secondary endpoints were prednisone dose required to control disease activity.
  The average daily dosage of prednisone that was employed to control disease activity was diminished from 24.3±4.7 mg/day upon enrollment at visit 1 to 7.2±2.3 mg/day upon termination of the 12-month treatment period at visit 6.
Time Frame: 1 year
Population: SLE patients
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SLE Subjects Receiving the Study Drug
Number analyzed (Participants) | 40
mg
  Prednisone dose upon enrollment at visit 1 | 24.3 (4.7)
  Prednisone dose upon termination of the 12-month treatment period at visit 6 | 7.2 (2.3)

ADVERSE EVENTS:
Groups:
- SLE Subjects Receiving the Study Drug: SLE Subjects receiving the study drug, Rapamune. Rapamycin: Rapamycin, is given to this group at a starting dose of 2 g/day
Arm/Group | SLE Subjects Receiving the Study Drug | Controls
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/56
Other Adverse Events (participants affected / at risk) | 1/40 | 0/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SLE Subjects Receiving the Study Drug (N=40) | Controls (N=56)
Oral ulcer (Gastrointestinal disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes